CLINICAL TRIAL: NCT01814709
Title: A Phase 1, Open-Label Study to Evaluate the Effect of Rifampin or Itraconazole on the Pharmacokinetics of GDC-0032 in Healthy Subjects
Brief Title: A Drug Interaction Study of GDC-0032 Co-administered With Rifampin or Itraconazole in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GP28617
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 2-(3-(2-(1-isopropyl-3-methyl-1H-1,2-4-triazol-5-yl)-5,6-dihydrobenzo(f)imidazo(1,2-d)(1,4)oxazepin-9-yl)-1H-pyrazol-1-yl)-2-methylpropanamide; Itraconazole; Rifampin

ARMS (2):
- Itraconazole Arm (Experimental)
  Interventions: Drug: GDC-0032; Drug: Itraconazole
- Rifampin Arm (Experimental)
  Interventions: Drug: GDC-0032; Drug: Rifampin

INTERVENTIONS:
Drug: GDC-0032 — Oral doses of GDC-0032
Drug: Itraconazole — Oral doses of Itraconazole
  Arms: Itraconazole Arm
Drug: Rifampin — Oral doses of Rifampin
  Arms: Rifampin Arm

SUMMARY:
This open-label, two-arm, drug interaction study will investigate the effect of co-administration of rifampin or itraconazole on the pharmacokinetics of GDC-0032 in healthy volunteers. In Arm A, volunteers will receive GDC-0032 and rifampin; in Arm B, volunteers will receive GDC-0032 and itraconazole. The anticipated time on study treatment is approximately 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Female volunteers will be non-pregnant, non-lactating, and either postmenopausal for at least 1 year or surgically sterile
* Male volunteers will either be sterile, or agree to use adequate methods of contraception
* Body mass index (BMI) range 18 to 32 kg/m2, inclusive
* No clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs; and clinical laboratory evaluations
* Negative hepatitis B virus, hepatitis C virus and negative HIV antibody screens

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* History of stomach or intestinal surgery or resection that would alter absorption and/or excretion of orally administered study drugs
* History of alcoholism or drug addiction within 1 year prior to Check-in
* History of chronic proton pump inhibitor (PPI) use within 6 months of Check-in, or use of PPIs, H2-receptor antagonists, or antacids within 1 month prior to Check-in and during the entire study
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* History type 1 or 2 diabetes and/or elevated fasting glucose at baseline
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Use of any tobacco- or nicotine containing- products
* Participation in any other investigational study drug or biologic agent trial in which receipt of an investigational study drug occurred within 5 half-lives or 30 days, whichever is longer to Check-in and during the entire study duration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Plasma concentrations of GDC-0032 | 2 months
Safety: Incidence of adverse events | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Dallas, Texas, United States